CLINICAL TRIAL: NCT05423678
Title: In Depth Observational Clinical Trial - Analyzing Participation Experiences Of Amyotrophic Lateral Sclerosis Patients
Brief Title: Clinical Trial - Analyzing Participation Experiences Of Amyotrophic Lateral Sclerosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12207799
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis
Keywords: als; als clinical trials; als diversity studies; amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trial participation has always been substantially skewed toward certain demographic groups. However, there has been little study on whether trial qualities impact participation in either a positive or negative way. The goal of this research is to identify the characteristics that consistently restrict patients' ability to participate in or complete a trial in which they were initially interested. This data will be analyzed via a number of demographic lenses in order to find trends that could benefit future ALS sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the United States
* Is 18+ years old
* Participant has a diagnosis of Amyotrophic Lateral Sclerosis (ALS)
* Participant has enrolled in an interventional clinical for ALS (self-reported)

Exclusion Criteria

* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form
* No diagnosis of Amyotrophic Lateral Sclerosis (ALS) confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Amyotrophic Lateral Sclerosis patients who are actively considering enrolling in an interventional clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patient decides to enroll in clinical trial | 3 months
Rate of patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chio A, Canosa A, Gallo S, Cammarosano S, Moglia C, Fuda G, Calvo A, Mora G; PARALS group. ALS clinical trials: do enrolled patients accurately represent the ALS population? Neurology. 2011 Oct 11;77(15):1432-7. doi: 10.1212/WNL.0b013e318232ab9b. Epub 2011 Sep 28. PMID 21956723
- [Background] Sabatelli M, Conte A, Zollino M. Clinical and genetic heterogeneity of amyotrophic lateral sclerosis. Clin Genet. 2013 May;83(5):408-16. doi: 10.1111/cge.12117. Epub 2013 Mar 12. PMID 23379621
- [Background] Powell JH, Fleming Y. Making medicines for America: the case for clinical trial diversity. J Natl Med Assoc. 2000 Nov;92(11):507-14. No abstract available. PMID 11152082

DOCUMENTS (1):
  • Informed Consent Form (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT05423678/ICF_000.pdf